CLINICAL TRIAL: NCT02982967
Title: The Impact of the Recreational Physical Activity on Irisin Levels, Endothelial Progenitor Cells and Metabolic Profile in Healthy Children
Brief Title: Recreational Physical Activity and Cardiometabolic Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Maria do Carmo Pinho Franco, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013/03139-0
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Physical Activity; Endothelial Dysfunction; Metabolic Syndrome x
Keywords: child; physical activity; irisin; EPCs
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical Activity (Other): Single-arm study with recreational physical activity intervention by 10 weeks (Duration: 60 minutes; Intensity: 65%-85% heart rate reserve; Frequency: 4 sessions/week).
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Physical Activity — Recreational Physical Activity (Duration: 60 minutes; Intensity: 65%-85% heart rate reserve; Frequency: 4 sessions/week).

SUMMARY:
The purpose of present study was to investigate the effect of 10 weeks of recreational physical activity program on the irisin levels, progenitor endothelial cells and cardiometabolic profile in healthy children. Also, we investigated the correlation between this markers with anthropometric data, body composition, cardiac autonomic balance and physical fitness parameters. We evaluated eighty children aged 6 to 14 participated in the recreational physical activity program by 10 weeks (Duration: 60 minutes; Intensity: 65%-85% heart rate reserve; Frequency: 4 sessions/week). All parameters were evaluated before and after this approach.

DETAILED DESCRIPTION:
This cross-sectional study was conducted in a representative group of children aged 6 to 14 identified in the Youth Healthcare Centre located near the Federal University of São Paulo (São Paulo, SP, Brazil). A total of 110 children were identified during the study period. However, five individuals with respiratory problems and 12 individuals who did not agree to participate were excluded from the study. In addition, 13 individuals who have not completed anthropometric, metabolic or physical fitness assessments in the post-training period were also excluded. Therefore, 80 children (32 girls and 48 boys) were included for this study. No child had any clinical signs of musculoskeletal or orthopedic disorders that prevented them from performing the proposed physical fitness tests. The Ethics Committee of the Federal University of São Paulo approved the study protocol (Number: 795.262). All parents and children signed written informed consent/assent forms.

Experimental Design: Each child completed the experimental protocol over a period of 10 weeks consisting of the baseline measurements of anthropometric data, body composition, irisin levels, metabolic and physical fitness parameters. All these measurements were repeated after the 10-week recreational physical activity program and were carried out within 72 hours after the last training session.

Recreational Physical Activity Program: Participants performed 10 weeks of recreational physical activity program on circuit training, that consists of exercise program for flexibility, coordination, strength (upper and lower limbs), aerobic resistance controlled by use of the Polar S810i monitor (Polar Electro OY, Finland; sampling rate=100Hz) and dynamic balance to improve the functional capacity. A total of 40 sessions were performed with duration (60 minutes), intensity (65%-85% heart rate reserve), and frequency (4 sessions/week). Each session consisted of three parts: Warm-up (10 minutes), physical activity session (45 minutes) and cool down (5 minutes). Moreover, subjective Borg scale of perceived exertion was applied to all children for control of the training intensity.

Anthropometry: Body weight and height were measured in light clothing without shoes using a standard balance beam scale. Waist and hip circumferences were measured using inextensible tape. Waist circumference was recorded at a level midway between the lower rib margin and the iliac crest at the end of normal expiration. .

Body Composition: Body composition was evaluated using bioelectrical impedance with a single-frequency hand-to-foot (ImpediMed DF50 monitor, Impedimed, Australia). Children were asked to avoid physical activity and to consume liquids 2 hours before evaluation to prevent errors in measurement due to fluid imbalances. This evaluation was performed after 5 minutes of rest in the supine position, and the electrodes were applied to the hand, wrist, ankle and foot of the right-hand side of the body. Body fat was calculated with prediction equations.

Cardiorespiratory Fitness: The 20-meter shuttle run test (20MST) was performed to estimated cardiorespiratory fitness. The test starts at 8 km/h and increases by 0.5 km/h every minute. This test was carried out in a plane surface, and explained by the field team member. All children made adaptations to the 20MST test. The velocity in the last stage completed by each child was recorded and used to calculate the VO2max (ml/kg/min) according to the equation proposed by Léger et al.

Standing Broad Jump: The child stands behind a line marked on the ground. A two foot take-off and landing is used, with swinging of the arms, the child jumps as far as possible with both feet simultaneously. The test item score (better of three attempts) is the distance between the starting line and the landing position (measured in centimeters).

Sit and Reach Test: The flexibility was evaluated by use of the Wells Bench. For this test, the child performed the movement with hands overlapped, feet rested on the bench and knees totally extended with aid from the researcher. The result was given by the maximum distance obtained in three attempts, respecting a one-minute interval between them.

Handgrip Strength Test: Grip strength was measured for both hands using a digital dynamometer (Kern & Sohn, Model MAP 80K1S, Germany). In this test, the child was seated in appropriately sized chairs, shoulder abducted, elbow in 90 degrees flexion, and wrist in neutral position. After that, the researcher asked the child to perform the greatest possible force in the shortest time. The mean of three maximum voluntary contractions was recorded for each hand and expressed in Kg.

Blood Collection and Biochemical Variables: In the morning (7:00 - 9: 00hrs) after overnight fasting, the blood venous samples (10 ml) were collected by venipuncture of a forearm vein into separate vacutainer tubes containing spray-dried K2EDTA anticoagulant or with gel serum separator. EDTA samples were centrifuged within 1 hour after blood collection (4°C - 1,500 g for 15 min) and plasma aliquots for irisin measurement were stored at -80°C until assay. Automated enzymatic procedures were used to measure glucose and insulin by routine methods in Clinical Laboratory of the Kidney & Hypertension Hospital. Insulin resistance was calculated by the homeostasis model assessment (HOMA-IR) method, according to the following formula: [glucose (mg/dl)/18 x insulin (mUI/ml)]/22.5.

Assessment of Irisin: Plasma irisin levels were determined using commercially available ELISA kit (MyBioSource, Catalog Number: MBS 706887, San Diego, CA, USA). The intra assay and inter assay coefficients of variation were less than 8%. These assays were performed in duplicate, and to remove any bias, the researcher devised blind analysis techniques.

Hemodynamic Variables and Heart Rate Variability: Blood pressure levels were measured twice in the right arm with the child in a seated position using an automated oscillometric device (Omron HEM907XL; Omron Healthcare; USA) with an appropriate cuff size. The blood pressure value was the average of three measurements made at 2-min intervals . After this procedure, children were asked to lay silently in a supine position on a bed with minimal body movement and to maintain spontaneous breathing for 10 minutes to record both resting heart rate and short-term heart rate variability using a Polar S810i monitor (Polar Electro OY, Finland; sampling rate=100Hz) . The same researcher blinded to the clinical data conducted the assessment of all children.

Processing of the Heart Rate Variability Data: The heart rate variability indices were calculated as previously described 27, 28. Briefly, normal beat to beat intervals were transferred from Polar S810i to Precision Performance Software by an infrared interface device. These data were processed in a specific previous routine designed in MatLab (Math Works, 6.0 version, USA) for the automatic selection of 5 minutes RR with the smallest variance. Afterwards, these time series lasting 5 minutes were analyzed in Kubios software (Biosignal Analysis and Medical Image Group, University of Kuopio, Finland). In this software, the artifacts were corrected with a moderated filter, and the time-domain components were calculated. The following time-domain indices were analyzed: heart rate (HR), MNN (average of all normal RR interval), SDNN (standard deviation of RR intervals), RMSSD (root mean square of successive differences RR intervals), and pNN50 (percent RR intervals with a difference in duration higher than 50 ms). The frequency-domain components were also evaluated by a 2 power spectrum. The classical frequency low frequency (LF= 0.041-0.15 Hz) and high frequency (HF= 0.15-0.40 Hz) bands were expressed in normalized units (n.u.). Moreover, the ratio of LF/HF was also calculated. Spectral analysis was estimated as recommended using the non-parametric method of fast Fourier Transform Algorithms.

Isolation of Peripheral Blood Mononuclear Cells: In this assay 5-6 mL from peripheral blood were collected in EDTA tubes. Under sterile conditions, tibia and femur cavities were flushed with DMEM (Dulbecco's Modified Eagle's medium, GIBCO, USA) to obtain bone marrow (BM). PB and BM were fractioned by gradient density centrifugation (2.500 rpm, 25 min, 20-22°C) (Ficoll-Paque, GE, Germany), and then, mononuclear cells obtained from its samples were addressed to number quantification and in vitro function.

Endothelial progenitor cells Immunophenotyping and Quantification by Flow Cytometer: mononuclear cells was considered endothelial progenitor cells as CD34+/VEGFR2+ cells. Briefly, 1x106 mononuclear cells were individually incubated (room temperature, in the dark, 30 min) with the following antibodies: anti-CD34-PeCY7 plus VEGFR2-FITC or with isotype controls anti-IgG-PE-Cy7 plus IgG-FITC . After incubation, cells were washed in PBS and fixed in 1% paraformaldehyde solution. Fixed cells were kept (4°C, in the dark, for 15-20 hours), and then analyzed in flow cytometer (FACSCANTO, BD Biosciences, USA) by collecting 1.000.000 events. Data were analyzed using BD FACSDIVA Software . Gates were established on the forward- and side-scatter (FSC/SSC) plot corresponding to select mononuclear cells followed by CD34-PeCY7 plus VEGFR2-FITC gate . Number of EPCs (CD34+/VEGFR2+) was calculated as the percentage of CMNs events30.

Endothelial progenitor cells - Functional Capacity in vitro Assay: Mononuclear cells were individually addressed to colony forming unit in vitro. Briefly, 5x106 MNCs were cultured (37°C, 5% CO2, 95% humidity) on 6-wells pre-coated fibronectin seeded with EndoCult medium . After 48 hours, 1x106 non-adherent cells were transferred in triplicate onto 24-wells pre-coated fibronectin and cultured for 72-96 hours (37°C, 5% CO2, 95% humidity) in EndoCult medium. Following, the colony forming units were counted manually by 2 blinded observers in inverted microscope.

Statistical Analysis: Statistical analyses were conducted using SPSS version 21.0 for Windows (IBM Corporation, USA). Categorical variables were compared using the chi-square test. All continuous variables were examined for normality with the Shapiro-Wilk test. Since our data had a nonparametric distribution was used Wilcoxon test for paired data in order to evaluate the difference between the baseline and post-Recreational physical activity program values. In addition, we used Spearman's rho correlation coefficient to determine the relationship between irisin and independent factors. The data were expressed as the mean ± standard deviation. Statistical tests were two-tailed and the significance level was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children
* Both Gender
* Aged 6 to 14 years

Exclusion Criteria:

* Clinical signs of musculoskeletal or orthopedic disorders that prevented them from performing the proposed physical fitness tests.
* Not completed anthropometric, metabolic or physical fitness assessments in the post-physical activity period

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
improvement in body composition | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria do Carmo Franco, PhD, Principal Investigator — Associate Professor
Locations (1):
- Physiology Department - Federal University of são Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Souza LV, De Meneck F, Fernandes T, Oliveira EM, Franco MDC. Physical activity intervention improved the number and functionality of endothelial progenitor cells in low birth weight children. Nutr Metab Cardiovasc Dis. 2020 Jan 3;30(1):60-70. doi: 10.1016/j.numecd.2019.08.011. Epub 2019 Aug 30. PMID 31753788
- Available data/document: Individual Participant Data Set — https://figshare.com/s/8f238bd02ca631cfe5fd